CLINICAL TRIAL: NCT00248209
Title: A Multi-center, Double-blind, Placebo-controlled Study of Bupropion XL in Females With Orgasmic Disorder
Brief Title: Female Orgasmic Disorder (FOD) and Wellbutrin XL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Segraves, R., T., M.D., Ph.D. (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Segraves, R.T. M.D., Ph.D, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GSK FOD
Record Dates: First submitted 2005-11-01; First posted 2005-11-03 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2007-04

CONDITIONS: Orgasmic Disorder
Keywords: Female Orgasmic Disorder; Female Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wellbutrin XL or placebo (Placebo Comparator): 1 arms - Wellbutrin XL or placebo
  Interventions: Drug: Wellbutrin XL

INTERVENTIONS:
Drug: Wellbutrin XL — Patients randomized to the bupropion treatment group will receive bupropion XL150 mg in the AM for 7 days increasing to 300mg/day (single daily dose). The investigator can increase the dose to 450mg per day at Day 28 if clinically indicated.
  Other Names: bupropion XL, Wellbutrin XL

SUMMARY:
A recently completed multi-site double-blind placebo-controlled study found that bupropion (Wellbutrin XL) increased female orgasmic function in a group of pre-menopausal women with a diagnosis of hypoactive sexual desire disorder. The purpose of this study is to ascertain whether bupropion will improve orgasmic function in pre-menopausal women with a primary complaint of idiopathic orgasmic disorder who do not have hypoactive sexual desire disorder. This will be a multicenter, placebo-controlled, double blind study of women with a diagnosis of female orgasm disorder. During a baseline visit, psychiatric, medical, alcohol and drug, and sexual histories will be obtained. Patients who continue to meet screening inclusion/exclusion criteria at their baseline visit will be randomly assigned to either placebo or bupropion XL for 8 weeks. A flexible dosing paradigm will be used. Sexual desire and activity will be assessed by patient diaries, investigator interview of sexual functioning every two weeks, and by standardized questionnaire every four weeks. The primary endpoint will be the increase in orgasm completion as measured by the Changes in Sexual Functioning Questionnaire-F (CSFQ-F). Secondary endpoints will be changes in sexual arousal, sexual desire, and sexual pleasure as assessed by the CSFQ-F.

DETAILED DESCRIPTION:
Background:

Female orgasmic disorder is characterized by a recurrent or persistent difficulty in achieving orgasm during sexual activity. A study of sexual activity in a representative sample of the US population ages 18-59 found that 24% of US females complained of significant difficulty achieving orgasm in the preceding year (Laumann et al, 2000). Epidemiological studies in Sweden and the United Kingdom have found similar rates of orgasm disorder.

Studies of drugs with actions of increasing genital vasodilation in response to sexual stimulation (eg alprostadil, sildenafil, or phentolamine) have generally been found to be unsuccessful or to have extremely limited efficacy in reversing female sexual dysfunction (Basson, 2001; Segraves, 2002). High doses of androgen have been shown to increase various parameters of sexual interest and activity in women after hysterectomy and bilateral oophorectomy (Schifren et al, 2000) and there is some evidence that oral dehydroepiandrosterone may increase responsiveness to sexual stimuli in postmenopausal women (Hackbert & Heiman, 2002).

There have been fewer studies of pharmacological treatment for hypoactive sexual desire disorder in premenopausal women. Extensive literature indicates that bupropion has a very low incidence of drug-induced sexual dysfunction (Clayton et al, 2002; Croft et al, 1999; Segraves & Balon, 2003) and that bupropion may reverse sexual dysfunction associated with serotonergic antidepressants (Rosen et al, 1999; Kennedy et al, 2002). In addition one controlled study (Crenshaw et al, 1987) and several clinical series indicate that bupropion may have prosexual effects in non-depressed females (Modell et al, 2000). A single blind study (Segraves et al, 2001) found that bupropion increased the frequency of episodes of sexual arousal and desire for sexual activity in women diagnosed with hypoactive sexual desire disorder.

A recent multicenter, double-blind, fixed dose study of females with global, acquired hypoactive sexual desire disorder found evidence that an exposure to 300 to 400 mg bupropion XL increased orgasm and pleasure as measured by the CSFQ-F. In this pilot study, all women had total serum testosterone levels within normal limits and were in stable, non-conflictual relationships. All patients had no evidence of psychiatric disorder and no evident etiology to their sexual complaint. All were pre-menopausal. The pilot study observed the effects of drug treatment for four months. Significant change in measures of sexual orgasm occurred as early as day 28. There are no currently approved pharmacological treatments for women with orgasmic disorder.

Specific Aims:

The purpose of this study is to delineate the effects of bupropion XL in women with global orgasmic disorder, using double blind conditions in an 8 week flexible dose multisite comparison of bupropion XL and placebo. It is hypothesized that bupropion XL will increase orgasm completion.

The primary objective of this study is to evaluate the effect of bupropion XL on the ease and frequency of achieving orgasm in sexual activity.

Secondary objectives will be to investigate the effects of bupropion XL on changes in sexual arousal and sexual pleasure.

ELIGIBILITY:
Inclusion Criteria:

A subject must:

1. Be able to understand and sign a written informed consent
2. Be a premenopausal female between 20 and 50 years of age, inclusive
3. Use active birth control, and be non-lactating, with a negative urine pregnancy test
4. Have no evidence of mood or anxiety disorder
5. Have a sexual partner who is without sexual dysfunction
6. Be in a stable, monogamous, sexual relationship of at least 6 months duration, and be willing to engage in sexual activity with a steady partner once a week for the duration of the study
7. Have no active psychiatric diagnosis
8. Have FOD which is not secondary to hypoactive sexual desire disorder or dyspareunia
9. Have English as first language or be fluent in English language
10. Meet operational definition of global female orgasmic disorder:

    1. Frequency of orgasm during sexual activity of less than 50% of sexual encounters
    2. Presence of disorder for at least six months
    3. At least 3 orgasms achieved in past 6 months
11. Have Beck Anxiety Disorder (BAI) scores less than 10
12. Have Beck Depression Inventory-II (BDI-II) scores less than 10
13. Have a CSFQ orgasm score of less than 11
14. Patient may have female arousal disorder as well as female orgasmic disorder

Exclusion Criteria:

1. Presence of organic condition known to cause sexual dysfunction (multiple sclerosis, diabetes mellitus, spinal cord injury)
2. Presence of hypoactive sexual desire disorder as defined below:

   1. Frequency of subjective sexual desire (interest in any type of sexual activity) less than or equal to once every two weeks
   2. Low intensity of sexual desire
   3. Frequency of self-initiated sexual activity less than or equal to once every two weeks
   4. Absence or low frequency of thoughts about sex (do not include thoughts of wishing for return of sexual interest): thoughts less than or equal to 4 times per month
   5. Presence of disorder for at least six months
   6. Absence of sexual desire includes all types of sexual activity
3. Taking psychiatric drugs other than study medication (zolpidem can be taken for a total of 10 days in trial for nighttime sedation)
4. Significant marital discord
5. Presence of sexual aversion disorder, dyspareunia, vaginismus, gender identity disorder, paraphilia
6. Drug or alcohol abuse in past year
7. History of seizure disorder or significant head injury
8. History of anorexia or bulimia
9. Taking any pharmacological agents known to be associated with sexual dysfunction (chronic opiate use, beta-blockers, alpha-adrenergic blockers, psychotropic medications)
10. Have an onset of orgasmic disorder within two months of beginning current hormonal contraceptive agent, if applicable
11. Have a cessation of menses for the three consecutive months prior to study entry
12. History of bilateral oophorectomy
13. Presence of dyspareunia

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2004-05; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the effect of bupropion XL on the ease and frequency of achieving orgasm in sexual activity. | 8 weeks of treatment

SECONDARY OUTCOMES:
Secondary objectives will be to investigate the effects of bupropion XL on changes in sexual arousal and sexual pleasure. | 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Segraves, MD, PhD, Principal Investigator — MetroHealth Medical Center/Case Western Reserve University
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States